CLINICAL TRIAL: NCT05565001
Title: Structural and Functional Cerebral Changes After Infusion of ATP Sensitive Potassium Channel Opener Levcromakalim.
Brief Title: The Involvement of ATP Sensitive Potassium Channel in Migraine Aura and Migraine Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, Study investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-21028500
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Headache; Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Headache; Migraine with Aura; Migraine without Aura | interventions — Cromakalim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator): Intravenous infusion of 1 mg levcromakalim followed by intravenous sumatriptan infusion.
  Interventions: Drug: Levcromakalim
- placebo (isotonic saline) (Placebo Comparator): Intravenous infusion of placebo (isotonic saline) followed by intravenous sumatriptan infusion.
  Interventions: Drug: Levcromakalim

INTERVENTIONS:
Drug: Levcromakalim — Intravenous administration of levcromakalim or placebo over 20 minutes. After 3 hours from the administration of levcromakalim or placebo, participants will receive intravenous infusion of sumatriptan over 10 minutes.

SUMMARY:
The aim of the present study to investigate whether

* Opening of KATP channels causes migraine pain by activation of meningeal nociceptors and ascending trigeminal nociceptive pathways.
* Opening of KATP channels causes migraine aura by induction of CSD.

DETAILED DESCRIPTION:
Migraine Pain The trigeminovascular system is the anatomical and physiological substrate of migraine pain. Nociceptive transmission originates from activation and sensitization of first-order trigeminovascular neurons. Their cell bodies are in the trigeminal ganglion, and their afferent fibers innervate the meninges and its vessels. Ascending nociceptive transmission from the trigeminal ganglion is projected to the brain stem, activating and sensitizing second-order trigeminovascular neurons, including those in the spinal trigeminal nucleus. This, in turn, activates and sensitizes third-order trigeminovascular neurons in the thalamus, which subsequently relay the nociceptive transmission to the somatosensory cortex and other cortical areas, ultimately resulting in migraine pain.

Although the biological underpinnings of migraine pain are incompletely understood, signaling pathways have been identified that are putatively responsible for the genesis of migraine pain. Recent human experimental data have implicated opening of KATP channels in migraine pathogenesis. In two randomized controlled trials, it was demonstrated that intravenous infusion of levcromakalim - an opener of KATP channels - induced migraine pain in people with migraine with and without aura.

- It remains unknown whether KATP channel opening causes migraine pain by activation of meningeal nociceptors and ascending trigeminal nociceptive pathways, as proposed during spontaneous migraine attacks.

Migraine Aura About one-third of people with migraine experience aura symptoms, which are characterized by reversible focal neurologic symptoms, typically comprising visual or hemisensory disturbances. The physiological substrate of the aura phase of migraine is thought to be cortical spreading depression (CSD), a self-propagating wave of depolarization across the cerebral cortex that disrupts ionic gradients and is followed by cerebral hypoperfusion. Recently, it was reported that intravenous infusion of levcromakalim - an opener of KATP channels - induced migraine aura in migraine with aura patients.

- It remains unknown whether KATP channel opening causes CSD which leads to migraine aura, as observed during spontaneous migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients
* 18-60 years.
* 50-100 kg.
* Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

* A history of serious somatic disease
* Any other type of headache (except episodic tension-type headache less than once a month) Daily intake of any medication except contraceptives Contraindications for MRI scan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic diffusion weighted image (DWI) | Before and after infusion of levcromakalim compared with before and after infusion of saline. Time of measurements is baseline, 20 minutes and 160 minutes after the infusion.
  To measure transient diffusivity changes related to levcromakalim-induced CSD during the aura phase of migraine in subjects with migraine with aura.

SECONDARY OUTCOMES:
Vascular imaging before sumatriptan | Before and after infusion of levcromakalim compared with before and after infusion of saline. Time of measurements is baseline, 20 minutes and 160 minutes after the infusion.
  To investigate the diameter of middle meningeal arteries (MMA), superficial temporal arteries (STA) and middle cerebral arteries (MCA) measured by millimeters (mm).
Vascular imaging after sumatriptan | Before and after infusion of sumatriptan. Time of measurements is 200 minutes and 210 minutes after the infusion.
  To investigate the diameter of middle meningeal arteries (MMA), superficial temporal arteries (STA) and middle cerebral arteries (MCA) measured by millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Danish headache center, Copenhagen, Glostrup, Denmark